CLINICAL TRIAL: NCT00621218
Title: A Pilot Study to Compare Tretinoin Gel, 0.05% to Tretinoin Gel Vehicle When Dosed Once or Twice Daily in Female Subjects With Classical Rosacea
Brief Title: A Study to Determine the Safety and Efficacy of Atralin (Tretinoin 0.05%) Gel for the Treatment of Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: D. Innes Cargill, PhD, Coria Laboratories, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9320-010-002
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Rosacea
Keywords: tretinoin, efficacy, safety, rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tretinoin gel 0.05%
- 2 (Placebo Comparator)
  Interventions: Drug: vehicle

INTERVENTIONS:
Drug: tretinoin gel 0.05% — Apply tretinoin gel, 0.05% topically once or twice daily to female subjects with rosacea
  Arms: 1
Drug: vehicle — Apply Atralin Gel vehicle topically once or twice daily to female subjects with rosacea.
  Arms: 2

SUMMARY:
To compare the efficacy and safety of tretinoin gel 0.05% to its vehicle when dosed once or twice daily in female subjects with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-65
* Diagnosed with classical, centrofacial, erythemato-telangiectatic rosacea

Exclusion Criteria:

* Male, females less than 18 years
* Females over 65 years
* No diagnosed rosacea

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Improvement in signs and symptoms of rosacea | 16 weeks

SECONDARY OUTCOMES:
Changes in various skin parameters | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Morris V Shelanski, MD, Principal Investigator
Locations (1):
- Product Investigations, Inc., Conshohocken, Pennsylvania, United States